CLINICAL TRIAL: NCT02479633
Title: Predetermınatıon of Root Coverage for Recessıons Treated wıth Coronally Advanced Flap wıth Connectıve Tissue Graft: An Exploratıve Study
Brief Title: Predetermination for Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Onur Ozcelik, Professor, Cukurova University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CukurovaU5
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Gingival Recessions
Keywords: prognostic factors
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- gingival recession type 1 (Other): recession defects without CAL intervention:Coronally advanced flap with connective tissue graft
  Interventions: Other: Coronally advanced flap with connective tissue graft
- gingival recession type 2 (Other): gingival recession with an amount of CAL equal or smaller to the buccal CAL. Intervention: Coronally advanced flap with connective tissue graft
  Interventions: Other: Coronally advanced flap with connective tissue graft

INTERVENTIONS:
Other: Coronally advanced flap with connective tissue graft — Two oblique, divergent releasing incisions extending beyond the mucogingival junction were performed. An intra-sulcular incision was performed at the buccal aspect of the involved tooth. Subsequently, a partial-thickness flap was raised beyond the MGJ. The papilla adjacent to the involved tooth were then de-epithelialized.
  The CTG was harvested using a single incision approach from the palate. The graft was positioned on the instrumented root surface immediately apical of the CEJ and then stabilized using a sling compressive crossing suture. The flap was coronally displaced 1-2 mm above the CEJ. A sling suture was placed to stabilize the flap in a coronal position, followed by interrupted sutures on the releasing incisions with an apico-coronal direction.
  Other Names: CAF+CTG

SUMMARY:
Background: The aim of present clinical study was to evaluate the predictive values of baseline inter-dental papilla height (IPH), avascular exposed root surface area (AERSA) and inter-dental clinical attachment loss (CAL) measurements on complete root coverage (CRC) of single gingival recession (GR) defects treated with coronally advanced flap and connective tissue graft technique (CAF+CTG).

Material and Methods: The study group included 65 females and 57 males, aged between 20 and 42 years. A total of 122 recession defects without CAL and with an amount of CAL equal or smaller to the buccal CAL , located at upper and lower incisors and canines were treated with CAF+CTG. IPH, AERSA and CAL parameters were analyzed for possible correlation with CRC after 6 months.

DETAILED DESCRIPTION:
The coronally advanced flap (CAF) with connective tissue graft (CTG) has been confirmed as the gold standard for treatment of gingival recessions ). CTG-based procedures provide the best outcomes with superior percentages of mean root coverage (MRC) and complete root coverage (CRC) and keratinized tissue (KT) gain. Data in previous reports show CRC range from 18% to 83% after CAF+CTG in Miller Classes I and II defects which are associated with no inter-dental clinical attachment loss (interdental-CAL) (Recession Type 1-RT1)

The use of CTG under CAF significantly enhances the probability to achieve CRC (%57) in recessions in which interdental-CAL is equal or smaller than the buccal attachment loss (Recession Type 2-RT2). It has been emphasized that CRC percentage was very similar to the result (60%) of a multicentre study on the treatment of RT1 recessions (Cortellini et al. 2009). Moreover, CRC was higher than most of the reports on treatment of RT1 or Miller I and II defects (more than 80%) when baseline interdental-CAL was between 1 and 3 mm Therefore, various CRC outcomes of the literature indicate that there is need for additional defect defining criteria for predicting the outcomes of root coverage (RC) in RT 1 and RT2 (interdental-CAL≤ 3mm) recession defects.

Predetermination of final RC which is important for distinguishing 'expected versus actual' amount of RC was found to be related to inter-dental papilla height (IPH) and inter-dental clinical attachment level (ICAL) by the clinical studies which reported correlation between these two anatomical characteristics and CRC. Recently a new predictive classification of gingival recessions using the baseline avascular exposed root surface area (AERSA) as an identification criterion has been proposed. AERSA resulted as a strong predictor of final RC after laterally positioned flap (LPF) leading to a prognostic model with AERSA explaining 86% of the mean root coverage. In addition, due to anatomic variations, some Miller Class I defects may have larger AERSA than Miller Class II and III defects or there may be smaller Miller Class III defects than Miller Class I and II defects which may significantly influence the treatment results. These results could help to explain the outcome variations among previous studies.

The prognostic anticipation of a certain amount of RC is a complex process including patient-related, tooth/site-related (GRD, root abrasion, ICAL, tooth type, the dimension of inter-dental papilla, AERSA) and technique-related (e.g. quality of the CTG) factors and operator's skill. It is essential to define the most potent prognostic factors' combination which can increase the success and predictability rates, to make CAF+CTG the most convenient RC technique for patients and clinicians. Therefore the aim of this study was to explore the predictive values of baseline IPH, AERSA and ICAL measurements on the final RC outcomes after CAF+CTG in RT1 and RT2 class GR defects.

ELIGIBILITY:
Inclusion Criteria:

* Presence of isolated RT1 and RT2 class gingival recessions with an AERSA ˃9mm2 on upper and lower incisors,
* Presence of identifiable cemento-enamel junction (CEJ); presence of a step ≤1mm at the CEJ level and/or the presence of a root abrasion, but with an identifiable CEJ,
* Full-mouth plaque score and Full-mouth bleeding score of <15%,
* No occlusal interferences;

Exclusion Criteria:

Exclusion criteria were:

* Patients with a history of periodontitis or abscess formation,
* Mucogingival or periodontal surgery at the experimental site in the last 1 year,
* Presence of systemic disease or taking medication known to interfere with periodontal tissue health,
* Smokers, pregnant patients.

Ages: 20 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
values of baseline interdental papill height | 1 year
  in mm

SECONDARY OUTCOMES:
avascular exposed root surface area | 1 year
  .n mm2
interdental clinical attachment level | 1 year
  in mm

CONTACTS AND LOCATIONS:
Overall Officials: Onur Ozcelik, Prof. Dr, Principal Investigator — Professor